CLINICAL TRIAL: NCT03651180
Title: Efficacy and Safety of Coronary Amphilimus-ELuting Stent in diAbeTic patiEnts: a Cross-sectional Multicentre Consecutive Study
Brief Title: Efficacy and Safety of Coronary Amphilimus-ELuting Stent in diAbeTic patiEnts
Acronym: ESCALATE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale S. Giovanni Bosco (Other)
Responsible Party: Principal Investigator, Salvatore Colangelo MD, Interventional Cardiologist, Ospedale S. Giovanni Bosco
Other Study IDs: 14942
Record Dates: First submitted 2018-05-10; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: Polymer free drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amphilimus eluting stent: Diabetic patients treated with Cre8 Amphilimus eluting stent
- Non Amphilimus eluting stent: Diabetic patients treated with any other drug eluting stent

SUMMARY:
More recently a polymer-free drug eluting stent (Amphilimus eluting stent) has shown to have a superiority in terms of efficacy and safety if compared with stable polymer drug eluting stent when used in diabetic patients. However, to date there are no direct comparisons of these two type of drug eluting stents.

DETAILED DESCRIPTION:
Drug eluting stent is the cornerstone of treatment in diabetic patients with coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI). However, there are a considerable number of patients who continue to have major adverse event despite this treatment. More recently a polymer-free drug eluting stent (Amphilimus eluting stent) has shown to have a superiority in terms of efficacy and safety if compared with stable polymer drug eluting stent when used in diabetic patients. These more favorable effects translate into reduced event rates, but to date there are no existing data comparing directly the mid-long term effect of this new polymer-free drug eluting stent with the other drug eluting stents in a larger cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of insulin or non-insulin dependent diabetes mellitus treated from at least 1 month
* if basal blood sugar at the admission is above 200 mg / dl or hemoglobin levels glycated> 6.5% (> 48 mmol / mol)

Exclusion Criteria:

* inability to provide informed consent or unable to guarantee the possibility of be contacted in the following 12 months;
* age under 18 years or over 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All diabetic patients undergone percutaneous coronary intervention with insertion of drug eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite endpoint of cardiac death, definite and probable stent thrombosis, re-PCI, Target Vessel Revascularization and bleeding in the two groups of study | 1 year
  Evaluation and comparison of the composite endpont of cardiac death, definite and probable stent thrombosis according with Academic Research Consortium criteria, Re-PCI, Target Vessel Revascularization, Type III and V bleeding complications according with Bleeding Academic Research Consortium criteria in the two groups of study

SECONDARY OUTCOMES:
Incidence of every single adverse event (cardiac death, definite and probable stent thrombosis, re-PCI, Target Vessel Revascularization and bleeding) in the two groups of study | 1 year
  Measurements and comparison of the incidence of any single adverse event of the composite endpoint (cardiac death, definite and probable stent thrombosis according with Academic Research Consortium criteria, Re-PCI, Target Vessel Revascularization, Type III and V bleeding complications according with Bleeding Academic Research Consortium criteria) in the two groups of study

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Colangelo, MD, Principal Investigator — San Giovanni Bosco Hospital - ASL Città di Torino
Locations (1):
- San Giovanni Bosco Hospital - ASL Città di Torino, Turin, Italy